CLINICAL TRIAL: NCT03978247
Title: Validation Study of the NASHMIR Test for Non-alcoholic Steatohepatitis (NASH) Diagnosis in Patients With Severe or Morbid Obesity
Brief Title: Signature Diagnostic of Non-alcoholic Steatohepatitis (NASH) by Infrared Light Spectroscopy
Acronym: SIGNALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diafir (Industry)
Collaborators: Clinact (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SIGNALS - 01; 2018-A03240-55 (Other: ANSM (ID-RCB))
Record Dates: First submitted 2019-04-23; First posted 2019-06-07 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The study is aimed at patients suffering from severe or morbid obesity and engaged in a bariatric surgery course. An additional blood sample will be taken upstream of the surgical procedure in the fasted subject. During the surgical procedure, a liver biopsy will be performed. The two diagnosis determined by the spectroscopic test and by means of the biopsy will then be compared to determine the diagnostic performance of the developped test (NASHMIR test).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NASHMIR group (Experimental): Validation of the NASHMIR Test
  Interventions: Diagnostic Test: NASHMIR

INTERVENTIONS:
Diagnostic Test: NASHMIR — An additional blood sample will be taken upstream of the surgical procedure and a liver biopsy will be performed in all included patients. The two results obtained by the spectroscopic test and by means of the biopsy will then be compared to determine the diagnostic performance of the developped test (NASHMIR test).

SUMMARY:
Evaluation of the diagnostic performance of an algorithm developed to detect metabolic profiles specific of non-alcoholic steatohepatitis NASH and based on the reading of a blood sample's infrared spectra

DETAILED DESCRIPTION:
The study is aimed at patients suffering from severe or morbid obesity and engaged in a bariatric surgery course. An additional blood sample will be taken upstream of the surgical procedure in the fasted subject. The metabolic fingerprint of the patient will be analyzed on serum from spectral data measured at most two hours after collection. The spectra obtained by the spectroscopy platform will be processed by algorithmic analysis to build the diagnostic test.

During the surgical procedure, a liver biopsy will be performed. The sample will be sent to the pathology laboratory for preparation and the slides will then be anonymized to be sent to a specialized laboratory for centralized reading by an expert pathologist. This expert will determine the diagnosis of non-alcoholic steatohepatitis (NASH) or non-NASH after microscopic analysis of the sample without having any information about the patient.

The two results obtained by the spectroscopic test and by means of the biopsy will then be compared to determine the diagnostic performance of the developped test (NASHMIR test).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old;
* Patient able to read, write and understand the French language;
* Patient who has signed an informed consent form before carrying out any procedure related to the study;
* Patient supported in bariatric surgery;
* Patient affiliated to a social security scheme or comparable scheme

Exclusion Criteria:

* Patient who has already benefited from a bariatric surgery (ring, sleeve, bypass ..);
* Patient taking: corticosteroid for more than 2 months, amiodarone, methotrexate, tamoxifen, 5-fluorouracil, irinotecan, cisplatin, asparaginase, nucleoside reverse transcriptase inhibitors of HIV, tetracycline, valproic acid, perhexilline;
* Patient with excessive alcohol consumption (> 210 g/week in men,> 140 g/week in women) present or past;
* Patient with infection or coinfection present or passed with hepatitis B virus, hepatitis C virus or human immunodeficiency virus;
* Patient with known chronic liver disease (including hemochromatosis, autoimmune hepatitis ...);
* pregnant, parturient or nursing women;
* Patient deprived of liberty by judicial or administrative decision;
* Patient subject to a legal protection measure;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance | 0-12 months
  The comparison of the results obtained by the mathematical analysis of the infrared spectra with those obtained by the reference method on histological samples from liver biopsies will allow to classify the results in true-positive, false-positive, true-negative and false-negative.
  The diagnostic performance of the signature will be evaluated by calculating the sensitivity, specificity, positive likelihood ratio, and negative likelihood ratio values.

SECONDARY OUTCOMES:
Diagnostic performance considering size | 0-12 months
  Diagnostic performance of the test taking into account size (cm). Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering current weight | 0-12 months
  Diagnostic performance of the test taking into account current weight (kg). Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering weight of the patient at the age of 20 | 0-12 months
  Diagnostic performance of the test taking into account Weight of the patient at the age of 20 (kg).
  Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering body mass index | 0-12 months
  Diagnostic performance of the test taking into account BMI (Body Mass Index) (kg/m2).
  Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering waist | 0-12 months
  Diagnostic performance of the test taking into account waist (cm). Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering hip circumference | 0-12 months
  Diagnostic performance of the test taking into account Hip circumference (cm). Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering systolic blood pressure | 0-12 months
  Diagnostic performance of the test taking into account systolic blood pressure (mmHg).
  Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering diastolic blood pressure | 0-12 months
  Diagnostic performance of the test taking into account diastolic blood pressure (mmHg).
  Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering type 2 diabetes | 0-12 months
  Diagnostic performance of the test taking into account type 2 diabetes (yes/No).
  Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering sleep apnea | 0-12 months
  Diagnostic performance of the test taking into account sleep apnea (Yes/No). Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering alcohol consumption | 0-12 months
  Diagnostic performance of the test taking into account current and/or previous alcohol consumption (Date and number of drinks per week).
  Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering tobacco consumption | 0-12 months
  Diagnostic performance of the test taking into account current and/or previous tobacco consumption (date and number of pack of cigarettes per year).
  Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering coffee consumption | 0-12 months
  Diagnostic performance of the test taking into account coffee consumption (number of cups per day).
  Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering cannabis consumption | 0-12 months
  Diagnostic performance of the test taking into account cannabis consumption (number of joints per week).
  Significance of each clinical parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant clinical variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the hemoglobin concentration | 0-12 months
  Diagnostic performance of the test taking into account the hemoglobin concentration (g/100mL).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the mean corpuscular volume | 0-12 months
  Diagnostic performance of the test taking into account mean corpuscular volume (fL).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the leukocyte count | 0-12 months
  Diagnostic performance of the test taking into account leukocyte count (Giga/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the platelet count | 0-12 months
  Diagnostic performance of the test taking into account platelet count (Giga/L). Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of aspartate transaminase | 0-12 months
  Diagnostic performance of the test taking into account aspartate transaminase (UI/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of alanine aminotransferase | 0-12 months
  Diagnostic performance of the test taking into account alanine aminotransferase (UI/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of gamma-glutamyl transferase | 0-12 months
  Diagnostic performance of the test taking into account the concentration of gamma-glutamyl transferase (UI/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of bilirubin | 0-12 months
  Diagnostic performance of the test taking into account the concentration of bilirubin (mg/dL).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of alkaline phosphatase | 0-12 months
  Diagnostic performance of the test taking into account the concentration of alkaline phosphatase (UI/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the prothrombin time | 0-12 months
  Diagnostic performance of the test taking into account the prothrombin time (%).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the blood glucose level | 0-12 months
  Diagnostic performance of the test taking into account the blood glucose level (mmol/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the HbA1c level | 0-12 months
  Diagnostic performance of the test taking into account the HbA1c level (hemoglobin A1c) (%).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of total cholesterol | 0-12 months
  Diagnostic performance of the test taking into account the concentration of total cholesterol (mmol/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of HDL cholesterol | 0-12 months
  Diagnostic performance of the test taking into account the concentration of HDL cholesterol (mmol/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of LDL cholesterol | 0-12 months
  Diagnostic performance of the test taking into account the concentration of LDL cholesterol (mmol/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of triglycerides | 0-12 months
  Diagnostic performance of the test taking into account the concentration of triglyceride (mmol/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of C reactive protein | 0-12 months
  Diagnostic performance of the test taking into account the concentration of C reactive protein (mg/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of ferritin | 0-12 months
  Diagnostic performance of the test taking into account the concentration of ferritin (g/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the concentration of albumin | 0-12 months
  Diagnostic performance of the test taking into account the concentration of albumin (g/L).
  Significance of each biological parameter will be assessed using statistical tests (mean comparison) on the two main populations (Non Alcoholic Steato Hepatitis Yes or No). Using logistic regression, a score calculated with significant biological variables will be aggregated to spectral score (primary outcome) in order to assess new diagnostic performance.
Diagnostic performance considering the subtype of non-alcoholic steatohepatitis determined through analysis of biopsy samples | 0-12 months
  Diagnostic performance of the test according to the different subtypes of non-alcoholic steatohepatitis (NAS score). NAFLD Activity Score calculated according to the steatosis grade (0, 1, 2 or 3), level of lobular inflammation (0, 1, 2 or 3) and stages of liver cell injury (0, 1 or 2)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolphe Anty, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Corvec M, Farrugia MA, Nguyen-Khac E, Regimbeau JM, Dharhri A, Chatelain D, Khamphommala L, Gautier AL, Le Berre N, Frey S, Bronowicki JP, Brunaud L, Marechal C, Blanchet MC, Frering V, Delwaide J, Kohnen L, Haumann A, Delvenne P, Sarfati-Lebreton M, Tariel H, Bernard J, Toullec A, Boursier J, Bedossa P, Gual P, Anty R, Iannelli A. Blood-based MASH diagnostic in candidates for bariatric surgery using mid-infrared spectroscopy: a European multicenter prospective study. Sci Rep. 2024 Nov 2;14(1):26452. doi: 10.1038/s41598-024-72704-5. PMID 39488538